CLINICAL TRIAL: NCT01765712
Title: "Effect of Intraoperative Application of Autologous PRP on Post Operative Morbidity in ACL Reconstruction Using Autologous Bone Patellar Tendon Bone Graft Harvest"
Brief Title: The Effect of Platelet Rich Plasma (PRP) on Post Operative Pain in Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brian Walters (Other)
Responsible Party: Sponsor-Investigator, Brian Walters, MD, Northwell Health
Organization: Northwell Health (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12-160A
Record Dates: First submitted 2013-01-03; First posted 2013-01-10 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Post Operative Pain
Keywords: PRP; BPTB; VAS; Anterior Knee Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Patients will be randomized into the treatment arm using a computer generated randomization table (simple randomization). Patients in the control arm of the study will undergo Anterior cruciate ligament reconstruction using Autologous bone patellar tendon bone autograft. At the end of the surgery, their graft donor site will have bone graft chips placed into the bony defect and the wound will be closed using sutures.
  Interventions: Procedure: Anterior Cruciate ligament reconstruction bone patellar tendon bone autograft
- Platelet Rich Plasma (Experimental): Patients randomized into the treatment arm of the study will undergo Anterior cruciate ligament reconstruction with Autologous bone patellar tendon bone autografts. At the start of the surgery,just after the administration of anesthesia, 10cc of blood will be withdrawn from the patients IV by the anesthesiologist. This sample will be spun down into 3-5cc of Platelet Rich Plasma which will be added to the patients bone graft chips and placed into the donor site at the end of the case.
  Interventions: Procedure: Anterior Cruciate ligament reconstruction bone patellar tendon bone autograft; Biological: Platelet Rich Plasma

INTERVENTIONS:
Procedure: Anterior Cruciate ligament reconstruction bone patellar tendon bone autograft
  Other Names: ACL; BPTB
Biological: Platelet Rich Plasma
  Other Names: PRP
  Arms: Platelet Rich Plasma

SUMMARY:
The purpose of this research study is to investigate whether or not platelet rich plasma (PRP) may help to improve tendon healing and decrease post operative pain in patients undergoing anterior cruciate ligament (ACL) reconstructive surgery using their own patellar tendons as autografts.

DETAILED DESCRIPTION:
There is currently a paucity of well-designed, prospective, randomized, blinded (Level 1) clinical studies that carefully and comprehensively investigate the role of PRP in ACL surgery. Specifically, ACL reconstruction using Bone Patellar Tendon Bone (BPTB) harvest and the role of PRP in decreasing postoperative pain at the donor site. Given the need for a highly powered study to demonstrate the clinical efficacy of PRP in ACL reconstruction, the investigators have designed a prospective, randomized, level 1, double-blinded study to evaluate the effects of PRP on the specific outcomes of donor site pain and radiographic measures of graft healing and incorporation.

The aim of this study is to evaluate the efficacy of intra-operatively applied autologous PRP in reducing donor site morbidity and increasing radiographic healing in ACL reconstruction using autologous BPTB.

ELIGIBILITY:
Inclusion Criteria:

* Primary ACL Reconstruction
* Outerbridge </= 2
* Minimum follow up of two years
* No ligamentous secondary injury
* Willingness to participate in study

Exclusion Criteria:

* Any previous knee injury
* prior history of anterior knee pain
* Outerbridge classification 3 or greater
* Revision ACL
* Diabetic or smoker
* Workers compensation patient
* pregnant or nursing women
* Any patient with limited English Proficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Nicholas, MD, Principal Investigator — Northwell Health
Locations (1):
- NY Orthopedics, New York, New York, United States

REFERENCES:
- [Derived] Walters BL, Porter DA, Hobart SJ, Bedford BB, Hogan DE, McHugh MM, Klein DA, Harousseau K, Nicholas SJ. Effect of Intraoperative Platelet-Rich Plasma Treatment on Postoperative Donor Site Knee Pain in Patellar Tendon Autograft Anterior Cruciate Ligament Reconstruction: A Double-Blind Randomized Controlled Trial. Am J Sports Med. 2018 Jul;46(8):1827-1835. doi: 10.1177/0363546518769295. Epub 2018 May 9. PMID 29741923

RESULTS

PARTICIPANT FLOW:
Groups:
- PRP Treatment: Patients treated with PRP
- Sham: Patients not receiving PRP
Period: Overall Study
Arm/Group | PRP Treatment | Sham
Started | 27 | 23
Completed | 27 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- PRP Treatment: 27 patients received the PRP treatment
- Sham Treatment: 23 patients received the sham treatment
- Total: Total of all reporting groups
Arm/Group | PRP Treatment | Sham Treatment | Total
Number analyzed (Participants) | 27 | 23 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 23 | 50
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (12) | 29 (12) | 30 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 28
  Male | 10 | 12 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 27 | 23 | 50

OUTCOME MEASURES:

1. Primary Outcome: Anterior Knee Pain
Description: The primary outcome measured will be anterior knee pain. The investigators will do so by using Visual Analog Scales as an assessment tool. The visual analog scales will include pain with activities of daily living and pain with kneeling activities. Information regarding these pain scales will be collected at 14 days and 1,3,6,12,18 and 24 months. The Visual analog Scale is a score from 0-10 with 0=no pain and 10=excruciating pain.
Time Frame: 2 weeks, 1, 3, 6, 12, 18, 24 months. Kneeling pain for treatment groups at 24 months post-op reported.
Population: Kneeling pain for treatment groups at 2 years post-op.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | PRP Treatment | Sham
Number analyzed (Participants) | 27 | 23
units on a scale | 2.4 (2.7) | 1.9 (1.6)
Statistical Analysis 1: Comparison: PRP Treatment vs Sham; Test type: Superiority; p = 0.55, t-test, 2 sided; Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-1.99 to 1.03]

2. Secondary Outcome: Radiographic Assessment of Tunnel Positioning
Description: A triple view radiographic series of the knee will be performed to assess the position of the tibial and femoral tunnels by one blinded senior radiologist.
Time Frame: 3 months
Population: Was not measured
Arm/Group | PRP Treatment | Sham
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Quantification of Healing at the Bony and Tendinous Harvest Sites
Description: Post-op MRI's will be obtained to quantify the amount of bony healing at the donor site and revascularization of native patellar tendon at the harvest site. These images will be interpreted by one blinded senior musculoskeletal radiologist.
Time Frame: 6 months
Population: MRI indices of donor site healing - defect in millimeters (mm)
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | PRP Treatment | Sham
Number analyzed (Participants) | 27 | 23
mm | 11.6 (2.4) | 12.0 (3.1)

4. Secondary Outcome: Post Operative Strength
Description: The objective clinical assessment of strength in the operative extremity will measured as quadriceps strength in a single leg hop test. This data will be collected by an independent researcher also blinded to treatment.
Time Frame: 3,6,12,18,24months
Population: Strength was not assessed
Arm/Group | PRP Treatment | Sham
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Post Operative Range of Motion
Description: The patients range of motion will be assessed on both the operative and non-operative knee. This information will be assessed using a goniometer and will be collected by a blinded clinician.
Time Frame: 2 weeks, 1,3,6,12,18,24months
Population: ROM was not measured
Arm/Group | PRP Treatment | Sham
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | PRP Treatment | Sham
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 0/27 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2012-09-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT01765712/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2014-05-14): https://cdn.clinicaltrials.gov/large-docs/12/NCT01765712/Prot_SAP_001.pdf